CLINICAL TRIAL: NCT02057926
Title: The Effect of Tetracycline in Degradation and Permeability of Collagen Membrane
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Mariana Baglivo, Periodontist, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C-45-ASA-08
Record Dates: First submitted 2014-01-22; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Ridge Preservation Technique
Keywords: Membrane degradation; Collagen membrane bio-durability
MeSH Terms: interventions — Metabolism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (1):
- Tetracycline, Without Tetracycline (Experimental): The study consist in two groups: test group (membrane treated with tetracycline) and control group (membrane no treated with tetracycline).
  Interventions: Drug: The effect of tetracycline in degradation and permeability of collagen membranes.

INTERVENTIONS:
Drug: The effect of tetracycline in degradation and permeability of collagen membranes.

SUMMARY:
The main objective of this study was to evaluate the histological impact of treatment with tetracycline (TTC) solution of two layers collagen membranes (CMs) bio-degradation, in ridge preservation technique (RPT). Additionally, secondary objectives were to evaluate the effect of TTC on bacterial colonization and inflammatory response. This is a randomized simple-blind clinical trial. Consecutive patients referred to the Department of Periodontology at Universitat Internacional de Catalunya (Barcelona, Spain), between November 2009 and April 2011, were included in the study. This study was based on data collected from 20 surgical sites in 10 systemically healthy patients requiring 2 extractions with SPT. Before starting the surgery, the two teeth of each selected patient were randomized in two groups. The test group underwent RPT with CMs embedded with TTC solution (CMs TTC), and the control group was performed without TTC solution (CMs NO TTC). Randomization was performed using SPSS software (version 18, SPSS Inc., Chicago, IL, USA). In the test group, both membranes were first dipped for 5 minutes in TTC solution (50 mg/ml). This involved the use of 250 mg tablets of TTC and 5 ml of saline that were mixed in a sterile trough. A sample of the membrane used in each SPT was retained as a negative control sample. The membrane sample was retrieved 7 days after initial surgery. At 14 days the suture was removed and a new control was performed within 1 month. A sample from the negative control, test and control group was analyzed from each patient. The specimens were fixed in a 10% formalin solution, dehydrated in a series of alcohols, embedded in paraffin, and sectioned in 4-5μ. The sections were stained with hematoxylin and eosin and examined with an Olympus BH-2 optical microscope. The stained sections were photographed with a digital camera mounted on an optical microscope at magnification (x100, x200 and x400). According to the findings of the present study, we can conclude that CMs exhibit rapid degradation when exposed to the oral environment. Histological interpretation suggests that CMs immersed in 50mg/ml TTC solution delay the CM degradation when exposed to the oral environment. Statistical evaluation did not show any difference in bacterial colonization and inflammatory response, but the findings may also be affected by the limited sample size.

The limits of the present study are the absence of histomorphometric analysis, the sample size, and the lack of a long-term evaluation with clinical evidence of the advantages of this technique. More clinical studies in humans are require to confirm the effect of TTC in CMs degradation before we can make recommendations.

ELIGIBILITY:
Inclusion Criteria: healthy patients with 2 teeth with hopless prognosis.

Exclusion Criteria: patients who had taken antibiotics 3 months prior to the study, patients with serious systemic disease, such as uncontrolled diabetes, cardiovascular disease and infectious diseases, patients that required antibiotic prophylaxis, patients who had received radiotherapy to the head and neck or chemotherapy in the past 12 months before treatment was proposed, untreated or uncontrolled periodontal disease, noncompliance with oral hygiene instructions, smokers of more than 10 cigarettes per day, pregnant women, patients allergic to tetracycline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the histological impact of treatment with tetracycline solution of two layers collagen membranes bio-degradation, in ridge preservation technique. | On week after surgery, a sample of the expose membrane was obtained. The sections were stained with hematoxylin and eosin and examined with an Olympus BH-2 optical microscope.
The main objective of this study was to evaluate the histological impact of treatment with tetracycline (TTC) solution of two layers collagen membranes (CMs) bio-degradation, in ridge preservation technique (RPT). | One week after the surgery, a sample of the expose membrane was obtained. The sections were stained with hematoxylin and eosin and examined with an Olympus BH-2 optical microscope.
  After 1 week, a sample of expose membrane was obtained. The bio-degradation of membrane was evaluated with a qualitative scale: 1) intact membrane, 2) partial degradation, 3) complete degradation.

SECONDARY OUTCOMES:
Secondary objectives were to evaluate the effect of tetracycline on bacterial colonization. | On week after surgery, a sample of expose membrane was obtained.The sections were stained with hematoxylin and eosin and examined with an Olympus BH-2 optical microscope.
  After 1 week, a sample of expose membrane was obtained. The bio-degradation of membrane was evaluated with a qualitative scale: 1) mild bacterial colonization, 2) moderate, 3) extensive.
Secondary objectives were to evaluate the effect of TTC on inflammatory response. | One week after surgery, a sample of exposure membrane was obtained. The sections were stained with hematoxylin and eosin and examined with an Olympus BH-2 optical microscope.
  After 1 week, a sample of expose membrane was obtained. The bio-degradation of membrane was evaluated with a qualitative scale: 1) absence of inflammatory response, 2) mild, 3) moderate, 4) marked.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Baglivo Duarte, Periodontist, Principal Investigator — Universitat Internacional de Catalunya; Antonio Santos, Periodontist, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat Del Vallès, Barcelona, Spain